CLINICAL TRIAL: NCT05084833
Title: ASPIRES (Activating Cancer Survivors and Their Primary Care Providers to Increase Colorectal Cancer Screening) Study
Acronym: ASPIRES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: St. Jude Children's Research Hospital (Other); Memorial Sloan Kettering Cancer Center (Other); Columbia University (Other); The Hospital for Sick Children (Other); Duke University (Other); Penn State University (Other); Hunter College of City University of New York (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000296; R01CA255269-01 (NIH)
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Early Detection of Cancer
Keywords: Colorectal cancer; cancer survivor
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group1: Control (C) (Experimental): Electronic educational materials (C).
  Interventions: Behavioral: Control
- Group 2: Patient Activation (PA) (Experimental): C + patient activation (PA) consisting of interactive tailored text messages with links to videos and resources
  Interventions: Behavioral: Control; Behavioral: Patient activation
- Group 3: Patient Activation and PCP Activation (PA + PCP) (Experimental): C + PA + PCP activation (PA+PCP) with physician materials about colorectal cancer risk in this population
  Interventions: Behavioral: Control; Behavioral: Patient activation; Behavioral: Primary care provider activation

INTERVENTIONS:
Behavioral: Control — Electronic educational materials
Behavioral: Patient activation — Interactive text messages with links to videos (e.g. colorectal cancer screening options, cost of colorectal cancer screening, perspective from a cancer survivor, why regular appointments are important for cancer survivors) and resources (e.g. helpful websites) are sent to participants
  Arms: Group 2: Patient Activation (PA); Group 3: Patient Activation and PCP Activation (PA + PCP)
Behavioral: Primary care provider activation — Faxed educational materials (e.g. current colorectal cancer screening recommendations, frequently asked questions, insurance letter template, cover letter with overview of patient's cancer treatment history) sent to primary care providers
  Arms: Group 3: Patient Activation and PCP Activation (PA + PCP)

SUMMARY:
The primary purpose of this study is to assess the best method for encouraging high-risk cancer survivors to get screened for colorectal cancer at the recommended age.

DETAILED DESCRIPTION:
This is a 12-month, 3-arm randomized controlled trial of 315 Childhood Cancer Survivor Study (CCSS) survivors using a text message intervention with data collected at baseline and 12 months through patient and provider surveys and interviews and a medical record review. Participants will be randomly assigned to one of three groups: control, patient activation (PA) using a text message/video intervention, or patient activation + primary care provider activation (PA + PCP) which will include providing primary care providers with resources about colorectal cancer risk in this population. All participants will receive electronic resources about their previous cancer treatment and colorectal cancer screening recommendations.

The primary outcome is the proportion of patients who complete the colonoscopy or Cologuard test (Cologuard test plus colonoscopy if the Cologuard is positive) within 12 months of enrolling on the study, as measured via self-report questions in the end of study questionnaire. The study will test the hypothesis that, compared to controls, survivors randomized to the PA and PA + PCP activation groups will have significantly higher rates of completion of colorectal cancer screening.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will include people who:

* Enrolled on the Childhood Cancer Survivor Study
* Were treated with radiation to the abdomen, pelvis, spine, or total body irradiation
* Have no history of colorectal cancer
* Have not had a colonoscopy in the last 5 years or Cologuard in the last 3 years
* Have a smartphone

Exclusion Criteria:

* Do not reside in the United States
* Do not speak English

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who report completing a colonoscopy or Cologuard test (Cologuard test plus colonoscopy if Cologuard is positive) within 12 months of randomization | 12 months
  This will be measured by self-report on a questionnaire given at 12 months.

SECONDARY OUTCOMES:
Proportion of patients who complete the colonoscopy or Cologuard test (Cologuard test plus colonoscopy if Cologuard is positive) within 12 months of randomization as measured in medical record reports | 12 months
  The study team will confirm if participants had a colonoscopy or cologuard test by reaching out to the medical site where the participant was screened, and requesting the medical record confirmation.
Potential barriers and facilitators to the uptake of the intervention at both the patient and provider level as measured by CFIR questions | 14 months
  Consolidated Framework for Implementation Research (CFIR) questions are included in the 12-month questionnaire for participants, the 12-month questionnaire for their primary care providers, and the end of study interviews for the participants, primary care providers, and other medical office staff. CFIR questions are meant to measure 5 domains: intervention characteristics, outer setting, inner setting, characteristics of individuals, and process.
Other potential barriers and facilitators to the uptake of the intervention at both the patient and provider level | 12 months
  In this study, the potential moderators include patient characteristics, such as age, gender, educational attainment, health insurance coverage, types of insurance, chronic health conditions, and race/ethnicity as well as PCP factors such as knowledge, years in practice, and practice setting. The potential mediators in this study may include the patient's perception of involvement in decision making, health insurance coverage, and whether the patient reviewed the study resources and videos. This will be measured through data collected via the baseline and 12 month questionnaires as well as data previously collected via the St. Jude Childhood Cancer Survivor Study.
Cost and Cost-Effectiveness Analysis | 12 months
  We will collect data on the replication costs of the intervention and health services from the intervention per participant. The costs of the intervention (e.g. intervention materials, personnel time, and texting costs) will be collected by the University of Chicago team via a cost spreadsheet. The cost of the health services will be collected via the 12-month questionnaire; participants will be asked to share information about the types of medical visits they have had since joining the study.

CONTACTS AND LOCATIONS:
Overall Officials: Tara O Henderson, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Karen Kim, MD, MS, Study Chair — The Pennsylvania State University
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University, New York, New York
  - The Pennsylvania State University, University Park, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No
Participants will be recruited from an established cohort (Childhood Cancer Survivor Study), and therefore individual participant data will not be available to other researchers.

REFERENCES:
- [Derived] Henderson TO, Bardwell JK, Moskowitz CS, McDonald A, Vukadinovich C, Lam H, Curry M, Oeffinger KC, Ford JS, Elkin EB, Nathan PC, Armstrong GT, Kim K. Implementing a mHealth intervention to increase colorectal cancer screening among high-risk cancer survivors treated with radiotherapy in the Childhood Cancer Survivor Study (CCSS). BMC Health Serv Res. 2022 May 23;22(1):691. doi: 10.1186/s12913-022-08082-3. PMID 35606736